CLINICAL TRIAL: NCT01560026
Title: Study for Elevate the Feasibility of Ovarian Preservation With Endometrial Carcinoma
Brief Title: Retrospective Study to Evaluate the Feasibility of Ovarian Preservation in Patients With Endometrial Carcinoma
Acronym: ECWOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Director, Taipei Veterans General Hospital, Taiwan
Other Study IDs: VHG0500
Record Dates: First submitted 2011-06-14; First posted 2012-03-21 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Endometrial Cancer
Keywords: ovarian preservation
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ovarian preservation: endometrial cancer with ovarian preservation
  Interventions: Procedure: surgery
- oophorectomy: endometrial cancer without ovarian preservation

INTERVENTIONS:
Procedure: surgery — endometrial cancer with or without oophorectomy
  Other Names: staging surgery with ovarian preservation
  Groups: ovarian preservation

SUMMARY:
Endometrial cancer is one of the most common female malignancies in the United States, and has increased in incidence in Taiwan in recent decades.A recent population-based analysis noted that 4% of endometrial cancers occurred in women aged 40 years or younger, furthermore it is up to 15% in Taiwan according to the data of cancer registry. The standard treatment of endometrial cancer results in surgical menopause and places patients at risk for the long-term sequelae of estrogen deprivation. The goal of this study was to determine the frequency of a coexisting ovarian malignancy and to evaluate the outcome of ovarian preservation in women with treatment for endometrial cancer.

DETAILED DESCRIPTION:
we reviewed the cases with early stage of endometrial cancer who have primary staging surgery between January 1989 to December 2009. The enrolled patients will be divided into two group (oophorectomy vs. ovary preservation) for analysis:the outcome and recurrence type.To evaluate the outcome of ovarian preservation in women with endometrial cancer .

ELIGIBILITY:
Inclusion Criteria:

* early stage endometrial cancer after primary surgery exclusion criteria:
* MMMT, type 2 endometrial cancer

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators retrospectively reviewed the cases of 150 patients who had primary surgery with early stage endometrial cancer between January 1989 and December 2009
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2000-08; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
from the time of diagnosis to the time of disease recurrence or last follow time | disease recurrence or last follow time, up to one year
  the time of diagnosis to the time of disease recurrence or last follow time

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, Study Chair — Department of Obstetric and Gynecology, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, ROC, Taiwan